CLINICAL TRIAL: NCT02647060
Title: The Exercise Capacity and Quality of Life in the Patients With Idiopathic Pulmonary Arterial Hypertension and Secondary Pulmonary Hypertension
Brief Title: The Exercise Capacity and Quality of Life in the Patients With IPAH and Secondary PH
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201511029RINA
Record Dates: First submitted 2015-12-15; First posted 2016-01-06 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Hypertension, Pulmonary
Keywords: cardiopulmonary exercise testing; right ventricle function; cardio output; pulmonary hypertension; quality of life
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- idiopathic pulmonary hypertension: 1. diagnose as idiopathic pulmonary arterial hypertension
  2. clinical stable over 3 months
  3. able to walk and can do bicycle cardiopulmonary exercise testing
- secondary pulmonary hypertension: 1. diagnose as pulmonary hypertension
  2. clinical stable over 3 months
  3. able to walk and can do bicycle cardiopulmonary exercise testing

SUMMARY:
Pulmonary hypertension (PH) is a progressive disease with high mortality rate, but due to the development of drugs, the prognosis of the disease has improved. However patients still have poor exercise capacity and decrease of the quality of life. Past studies have shown that idiopathic and secondary PH are different in etiology and prognosis. It is necessary to further understand the difference between exercise capacity and quality of life of these two types of patients.

DETAILED DESCRIPTION:
Background. Pulmonary hypertension (PH) is a progressive disease with high mortality rate, but due to the development of drugs, the prognosis of the disease has improved. However patients still have poor exercise capacity and decrease of the quality of life. Past studies have shown that idiopathic and secondary PH are different in etiology and prognosis. It is necessary to further understand the difference between exercise capacity and quality of life of these two types of patients.

Purpose. The purpose of this study is the comparison of idiopathic and secondary PH in exercise capacity and quality of life, and analyzed the factors affecting.

Method. The patients recruit from National Taiwan University hospital. Thirty patients who diagnosis with PH and willing to participant our study will recruited. According to the cause of disease patients will divided into two groups, idiopathic group and secondary PH group has fifteen patients. Both of group receive testing, including body composition, exercise capacity (six minutes walk test, cardiopulmonary exercise testing), record their regular physical activity( seven day physical activity recall questionnaire) , fatigue severity(fatigue severity scale), and quality of life (SF-36), monitor cardiac function (non-invasive cardiac output test instrument). Data are analyze using SPSS19.0 version. Data will be presented in mean ± standard deviation and percentage. Using Kolmogorov-Smirmov test to test, whether the data were normal distribution, when P> 0.05 is considered as a normal distribution. Mann-Whitney U test or Chi-square test to processing parameters between two groups. Independent sample t test will be used to compare whether there are between-group differences. Pearson correlation coefficient will be used to test correlations between the parameters. The study defines significant level at α = 0.05, two-tailed.

ELIGIBILITY:
inclusion criteria

1. diagnose as pulmonary hypertension
2. clinical stable over 3 months
3. able to walk and can perform cardiopulmonary exercise testing by bicycle

exclusion criteria

1. acute right heart failure
2. sever arrythmia
3. the history of exercise induce syncope

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pulmonary hypertension, clinical stable, able to walk and can perform cardiopulmonary exercise testing by bicycle
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-11-19 (Actual)

PRIMARY OUTCOMES:
exercise capacity | within 1 months after inclusion
  cardiopulmonary exercise testing(using ''MetaMax 3B system, CORTEX Biophysik GmbH'' as the measure system, and the data will present as VO2)
quality of life | within 1 months after inclusion
  SF-36
Functional exercise capacity | within 1 months after inclusion
  six minutes walk test

SECONDARY OUTCOMES:
Cardiac function | within 1 months after inclusion
  using non-invasive cardiac output test instrument (Bioelectrical impedance, Physioflow lab1), the data will present as cardiac output(CO)
Volume of regular physical activity | within 1 months after inclusion
  using "Seven day physical activity recall questionnaire"
fatigue severity | within 1 months after inclusion
  using "Fatigue severity scale"
body composition | within 1 months after inclusion
  using bioelectrical impedance (Maltron BioScan BF-920), the data will present as fat percentage

CONTACTS AND LOCATIONS:
Overall Officials: Chien Meng-Yueh, PhD, Study Director — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan